CLINICAL TRIAL: NCT01272089
Title: A Multi-Site, Open-Label Study of Patient Perception and Quality of Life Associated With the Use of Olopatadine 0.2% in Subjects With Allergic Conjunctivitis
Brief Title: A Study of Patient Perception and Quality of Life Associated With the Use of Olopatadine 0.2% in Subjects With Allergic Conjunctivitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-11-013
Record Dates: First submitted 2011-01-05; First posted 2011-01-07 (Estimated); Last update posted 2012-09-18 (Estimated); Status verified 2012-09

CONDITIONS: Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — Olopatadine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pataday (Experimental): Olopatadine Hydrochloride Ophthalmic Solution, 0.2%, one drop once daily for one week
  Interventions: Drug: Olopatadine Hydrochloride Ophthalmic Solution, 0.2%

INTERVENTIONS:
Drug: Olopatadine Hydrochloride Ophthalmic Solution, 0.2% — Olopatadine Hydrochloride Ophthalmic Solution, 0.2%, one drop once a day for one week
  Other Names: Pataday

SUMMARY:
The purpose of this study was to evaluate subject perceptions of Olopatadine 0.2%, dosed once-daily, in subjects with allergic conjunctivitis and to record any adverse events as described by the subjects as a part of this post marketing surveillance study.

ELIGIBILITY:
Inclusion Criteria:

* History (within the past 24 months) of allergic conjunctivitis.
* Willing to avoid contact lens wear for each of the study visits, immediately prior to study medication installation and for 10 minutes after installation of study drug.
* Contact lens wear should be stable and consistent for 3 months prior to Screening Visit (Day 1).
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Contraindications or hypersensitivity to the use of the study medication or its components.
* Inability or unwillingness to follow all study instructions and complete study visits as required.
* Subjects with only one sighted eye or not correctable (using ETDRS chart) to 0.6 log MAR or better in both eyes at the Screening Visit.
* A known history of recurrent corneal erosion syndrome (idiopathic or secondary to dry eye).
* Ocular trauma within six months prior to Visit 1 in either eye as determined by subject history and/or examination.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2011-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Overall Patient Satisfaction | Day 7
  As assessed by the subject on a questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Kolkata, India